CLINICAL TRIAL: NCT01670227
Title: Preventing Conduct Problems in Poor Urban Preschoolers
Brief Title: ParentCorps: Promoting Healthy Development in Children From Low Income Communities
Acronym: ParentCorps
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); U.S. Department of Education (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 5R01MH77331-2; R01MH077331 (NIH); R305F050245 (Other Grant/Funding Number: U.S. Department of Education)
Record Dates: First submitted 2012-08-08; First posted 2012-08-22 (Estimated); Last update posted 2023-06-15 (Actual); Status verified 2016-03

CONDITIONS: Behavior Problems of Childhood and Adolescence
Keywords: EARLY CHILDHOOD; UNIVERSAL PREVENTION

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- PARENTCORPS (Experimental): ParentCorps is a school-based, family-focused universal intervention designed to attenuate the multiple risks associated with urban poverty, on children's health and development
  Interventions: Behavioral: PARENTCORPS
- Control Condition (Other): No intervention
  Interventions: Behavioral: PARENTCORPS

INTERVENTIONS:
Behavioral: PARENTCORPS — ParentCorps is a culturally-informed, universal intervention (for all children enrolled in Pre-K within an elementary school) designed to promote positive behavioral supports for children at home and in the classroom. ParentCorps includes two complementary components: 1) parent and child group intervention (13 2-hour sessions after school) for Pre-K students and their families; 2) professional development and individual consultation for early childhood teachers.

SUMMARY:
The purpose of this study was to determine whether ParentCorps promotes academic achievement and prevents mental health problems in children living in disadvantaged urban communities

ELIGIBILITY:
Inclusion Criteria:

* Enrollment in Pre-K
* At least one English-Speaking caregiver

Exclusion Criteria:

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1050 (Actual)
Dates: Start 2005-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Academic achievement through Year 4 | Assessed twice per year in Years 1 and 2, and then annually through Year 4
  Academic achievement test scores assessed via the Kaufman Test of Educational Achievement (KTEA)
Change from baseline in Child behavior at school through Year 4 | Assessed twice per year in Years 1 and 2, and then annually through Year 6
  Masked observations of child behavior at school

SECONDARY OUTCOMES:
Change from baseline Academic performance through Year 4 | Assessed twice per year in Years 1 and 2, and then annually through Year 6
  Teacher and parent ratings of academic performance
Change from baseline Behavior through Year 4 | Assessed twice per year in Years 1 and 2, and then annually through Year 6
  Teacher and parent ratings of behavior
Change from baseline Parent engagement in school through Year 4 | Assessed twice per year in Years 1 and 2, and then annually through Year 6
  Teacher rating of parent engagement in school
Change from baseline Positive behavior support through Year 4 | Assessed twice per year in Years 1 and 2
  Parent report of positive behavior support
Change from baseline Classroom climate and positive behavior support through Year 4 | Assessed twice per year in Years 1 and 2, and then annually through Year 4
  Masked observations of classroom climate and positive behavior support

CONTACTS AND LOCATIONS:
Overall Officials: Laurie Brotman, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, The Child Study Center, New York, New York, United States

REFERENCES:
- [Background] Brotman LM, Calzada E, Huang KY, Kingston S, Dawson-McClure S, Kamboukos D, Rosenfelt A, Schwab A, Petkova E. Promoting effective parenting practices and preventing child behavior problems in school among ethnically diverse families from underserved, urban communities. Child Dev. 2011 Jan-Feb;82(1):258-76. doi: 10.1111/j.1467-8624.2010.01554.x. PMID 21291441
- [Result] Brotman LM, Dawson-McClure S, Huang KY, Theise R, Kamboukos D, Wang J, Petkova E, Ogedegbe G. Early childhood family intervention and long-term obesity prevention among high-risk minority youth. Pediatrics. 2012 Mar;129(3):e621-8. doi: 10.1542/peds.2011-1568. Epub 2012 Feb 6. PMID 22311988
- [Derived] Brotman LM, Dawson-McClure S, Kamboukos D, Huang KY, Calzada EJ, Goldfeld K, Petkova E. Effects of ParentCorps in Prekindergarten on Child Mental Health and Academic Performance: Follow-up of a Randomized Clinical Trial Through 8 Years of Age. JAMA Pediatr. 2016 Dec 1;170(12):1149-1155. doi: 10.1001/jamapediatrics.2016.1891. PMID 27695851
- [Derived] Brotman LM, Dawson-McClure S, Calzada EJ, Huang KY, Kamboukos D, Palamar JJ, Petkova E. Cluster (school) RCT of ParentCorps: impact on kindergarten academic achievement. Pediatrics. 2013 May;131(5):e1521-9. doi: 10.1542/peds.2012-2632. Epub 2013 Apr 15. PMID 23589806